CLINICAL TRIAL: NCT01148420
Title: Pilot Trial of Use of DMPA Injection and High Dose MPA Tablets in Outpatient
Brief Title: DMPA & High Dose Oral Progestin (MPA) Tablets in Outpatient Treatment of Acute Excessive Vaginal Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Women's Health Care Clinic, Torrance, California (Other)
Responsible Party: Principal Investigator, Anita Nelson, Medical Director, Women's Health Care Clinic, Torrance, California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13530-01
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Dysfunctional Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DMPA & MPA (Experimental): 150 mg intramuscularly received DMPA and two 10 mg tablets of MPA every 8 hours for 3 days
  Interventions: Drug: Medroxyprogesterone 17-Acetate; Drug: medroxyprogesterone acetate

INTERVENTIONS:
Drug: Medroxyprogesterone 17-Acetate — Medroxyprogesterone 20mg orally 3 times a day for 3 days
  Other Names: Provera; Cycrin
Drug: medroxyprogesterone acetate — Depo Provera 150mg Intramuscular injection
  Other Names: Depo Provera Injection

SUMMARY:
The purpose of this study is to investigate the effectiveness and acceptability of high dose MPA (20mg oral 3 times a day) for 3 days combined with an injection of DMPA 150 mg intramuscularly in the treatment of acute heavy, prolonged uterine bleeding who have been identified as being eligible for outpatient management

DETAILED DESCRIPTION:
Excessive vaginal bleeding is a frequent problem for reproductive age women and accounts for many office and emergency room visits. This bleeding is caused by cancer, endocrinologic problems, liver failure, benign tumors of the uterus, and cervix, as well as hormone imbalances, such as anovulatory cycling.

Even though excessive vaginal bleeding is very common, there has been very little research into ways to manage it. For non-pregnant women who have stable vital signs and are not hemorrhaging or experiencing severe anemia, outpatient therapy is generally attempted. Textbooks recommend treatment with high dose oral contraceptives pills (one tablet orally 2 times a day for 5 days). Recently, Munro et al published a small study using high doses of oral progestin (MPA 20mg 3 times daily for 7 days then one daily for 21 days). The median time to bleeding cessation was 3 days. Munro reported having difficulty enrolling adequate numbers of patients to achieve the statistical significance.

The investigators propose a pilot project to study clinical responses to a new hormonal therapy the blends the high dose oral therapy with the longer acting injectable progestin. The pilot clinical trial is designed to study 50 women who are bleeding and whose treatment is amenable to outpatient therapy. Routine care will be provided to each of the women before she is approached for study enrollment.

This study, therefore, is designed to provide short term proven therapy of 20 mg MPA tablets 3 times a day for 3 days combined with the injectable progestin (DMPA) that lasts for 3 months.

Patients will be called within 24 hours and 48 hours following their first study visit to ascertain their bleeding status and their use of medication, as well as any significant side effects they may be experiencing. Patients will be asked to return to the clinic on day 3 for a repeat hemoglobin and interval history. Those women who are still having any bleeding on day 3 will be contacted on day 5.

The primary outcome measures of the part of the study will be the time elapsed to slowing acute bleeding as well as compliance with study medications. The patient's time to complete cessation of bleeding and percent of women having complete bleeding cessation will also be calculated. Results of the biopsies done before randomization will also be evaluated to see if they had any influence on study outcomes. From the degree of responses seen in this pilot study, a larger clinical trial may be designed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 50
* Non-pregnant
* Candidate for outpatient management
* Able to understand and follow instructions
* Vital signs stable
* No severe anemia
* No medical conditions requiring transfusion

Exclusion Criteria:

* Pregnancy
* Breast cancer current or in last 5 years
* Allergy to MPA or DMPA
* Previous hormonal therapies
* Unstable vital signs
* Bleeding excessive enough to require surgical therapy or hospital admission
* Desire for pregnancy in next 6 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita L. Nelson, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Harbor-UCLA Urgent Care, Torrance, California, United States

REFERENCES:
- [Background] Speroff L, Fritz MA. Clinical Gynecologic Endocrinology and Infertility, 7th ed. Philadelphia: Lippincott Williams & Wilkins, 2005
- [Background] Munro MG, Mainor N, Basu R, Brisinger M, Barreda L. Oral medroxyprogesterone acetate and combination oral contraceptives for acute uterine bleeding: a randomized controlled trial. Obstet Gynecol. 2006 Oct;108(4):924-9. doi: 10.1097/01.AOG.0000238343.62063.22. PMID 17012455
- [Background] Munro MG, New Concepts in nongestational acute uterine bleeding.Contemporary Ob-GYN;53(1):52-57

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the GYN clinic at the Harbor-UCLA Medical Center.
Pre-assignment Details: Women were excluded if they were pregnant, hemodynamically unstable, had a known endometrial or cervical carcinoma, required immediate surgery, had hemoglobin less than 8, or had failed an earlier hormonal treatment for the current episode of bleeding.
Groups:
- DMPA + MPA: 150 mg intramuscularly received DMPA and two 10 mg tablets of MPA every 8 hours for 3 days.
Period: Overall Study
Arm/Group | DMPA + MPA
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DMPA + MPA
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 48
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.9 (8.09)
Hemoglobin baseline [Mean (Standard Deviation); unit: g/dL] | 10.9 (1.58)

OUTCOME MEASURES:

1. Secondary Outcome: Patient Perception of the Acceptability of the Treatment
Description: Results from a survey question that assessed the subjects' satisfaction with the therapy on a scale of 1-3. 1 = poor; 2 = good; 3 = excellent.
Time Frame: End of the trial; up to day 5
Measure: Median (Full Range); unit: units on a scale
Arm/Group | DMPA + MPA
Number analyzed (Participants) | 48
units on a scale | 3 [2 to 3]

2. Secondary Outcome: Satisfaction and Willingness to Recommend Treatment
Description: Participants were asked whether they would recommend this treatment to a friend
Time Frame: End of the trial; up to day 5
Measure: Number; unit: participants
Arm/Group | DMPA + MPA
Number analyzed (Participants) | 48
participants
  Participants who would recommend this treatment | 48
  Participants who would not recommend it | 0

3. Primary Outcome: Cessation of Bleeding Within 5 Days
Description: Patients were called within 24 hours and 48 hours following their first study visit to ascertain their bleeding status and their use of medication, as well as any significant side effects they msy have been experiencing. Patients were asked to return to the clinic on day 3 for a repeat hemoglobin and interval history. Those women who were still having any bleeding on day 3 were contacted on day 5
Time Frame: 3-5 days
Measure: Number; unit: participants
Arm/Group | DMPA + MPA
Number analyzed (Participants) | 48
participants | 48

ADVERSE EVENTS:
Time Frame: Five days
Groups:
- DMPA & High Dose MPA: DMPA & High Dose MPA
Arm/Group | DMPA & High Dose MPA
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 15/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DMPA & High Dose MPA (N=48)
Bloating (Reproductive system and breast disorders) | 7 — Potentially attributable to bleeding or anemia rather than to study medication.
Fatigue (Reproductive system and breast disorders) | 6 — Potentially attributable to bleeding or anemia rather than to study medication.
Cramping (Reproductive system and breast disorders) | 3 — Potentially attributable to bleeding or anemia rather than to study medication.
Mood changes (Reproductive system and breast disorders) | 2 — Potentially attributable to bleeding or anemia rather than to study medication.
Nausea (Reproductive system and breast disorders) | 1 — Potentially attributable to bleeding or anemia rather than to study medication.
Increased appetite (Reproductive system and breast disorders) | 1 — Potentially attributable to bleeding or anemia rather than to study medication.
Bone Pain (Reproductive system and breast disorders) | 1 — Potentially attributable to bleeding or anemia rather than to study medication.

LIMITATIONS AND CAVEATS:
This was a single-arm, noncomparative pilot clinical trial. Impacts on bleeding beyond 5 days were not prospectively documented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No